CLINICAL TRIAL: NCT00753870
Title: Range of Neutrophil Response to 20,000 EU of Clinical Center Reference Endotoxin in Otherwise Healthy Smokers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: David B. Peden, MD, MS, UNC_Chapel Hill
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07-2060 (GCRC 2670); P50HL084934-01 (NIH)
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Healthy Smokers
Keywords: current; no health problems; no daily cough from smoking
MeSH Terms: interventions — Lipopolysaccharides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Otherwise healthy smokers
  Interventions: Biological: CCRE inhalation

INTERVENTIONS:
Biological: CCRE inhalation — 20,000 EU CCRE given as a one-time challenge
  Other Names: CCRE (LPS)

SUMMARY:
Endotoxin is a component of outdoor air pollution, an air contaminant found in a number of different workplaces, and is even found in homes. The endotoxin used for this study is obtained from the National Institutes of Health, and is called "Clinical Center Reference Endotoxin", or CCRE. The purpose of this Phase 1 research study is to identify a dose of inhaled endotoxin that is safe (does not cause prolonged cough, shortness of breath or other problems), but causes changes in sputum cell samples that the scientists can measure. Phase 1 research studies like this one are not intended to be a treatment, but are a scientific investigation. Eventually, with these types of studies we will be able to examine why some people are more sensitive to endotoxin. Scientists at other universities have found that while most people do not have a considerable lung response to endotoxin at doses as high as 60,000 EU (endotoxin units), a few respond to as little as a total dose of 4500 EU. Our study is designed to identify if using a dose of 20,000 EU causes changes in the lung cells but does not cause symptoms in our study subjects. In our previous studies in our lab, using an endotoxin from another source, we have used higher doses (15,000 EUs) in subjects with asthma with no major problems, and we have used 10,000 EUs of CCRE in subjects who are current smokers without seeing any problems.

DETAILED DESCRIPTION:
We are looking for people who currently smoke a minimum of a half a pack of cigarettes each day. You must not have any other health problems, be pregnant or nursing a baby, or actively trying to become pregnant or to father a child.

ELIGIBILITY:
Inclusion Criteria:

* current smoker
* healthy

Exclusion Criteria:

* no asthma
* no chronic health conditions
* no daily cough
* not pregnant or nursing a baby
* not actively trying to get pregnant or father a child

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-08; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To identify a dose of inhaled CCRE that is well tolerated and that induces measurable increases in neutrophil content of induced sputum that can be employed to screen large populations for susceptibility to the inflammatory effect of inhaled endotoxin. | post exposure

CONTACTS AND LOCATIONS:
Overall Officials: David B Peden, MD, MS, Principal Investigator — University of North Carolina
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Bennett WD, Alexis NE, Almond M, Herbst M, Zeman KL, Peden DB. Effect of inhaled endotoxin on mucociliary clearance and airway inflammation in mild smokers and nonsmokers. J Aerosol Med Pulm Drug Deliv. 2014 Dec;27(6):459-65. doi: 10.1089/jamp.2013.1089. PMID 24568613
- See also: Related Info — http://www.med.unc.edu/cemalb/